CLINICAL TRIAL: NCT04137432
Title: Effects of an Oxytocin-augmented Cognitive-behavioral Group-based Short-term Intervention on Neural and Behavioral Correlates of Loneliness
Brief Title: Oxytocin-augmented Cognitive-behavioral Group-based Short-term Intervention for Loneliness
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University Hospital, Bonn (Other)
Collaborators: The German-Israeli Foundation for Scientific Research and Development (Other); Prof. Simone Shamay-Tsoory, University of Haifa (Unknown)
Responsible Party: Principal Investigator, Rene Hurlemann, Professor for Psychiatry, University of Oldenburg
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: GIF2
Record Dates: First submitted 2019-10-09; First posted 2019-10-24 (Actual); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Loneliness
Keywords: loneliness; oxytocin-augmented intervention; fMRI

STUDY DESIGN:
Intervention Model Description: Participants will receive either 24 IU of intranasal OT or placebo (PLC) over the four intervention sessions. All participants in one intervention group will receive the same substance.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxytocin (24 IU) (Experimental): Intranasal administration of 24 international units (IU) of oxytocin (OT) 30 minutes before the start of four intervention sessions
  Interventions: Drug: Oxytocin nasal spray
- Placebo (Placebo Comparator): Intranasal administration of a placebo spray 30 minutes before the start of four intervention sessions
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin nasal spray — Intranasal administration of 24 international units oxytocin.
  Arms: Oxytocin (24 IU)
Drug: Placebo — The placebo nasal sprays contains identical ingredients except for the peptide itself.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the clinical potential of oxytocin (OT) as an adjunct to a cognitive-behavioral group-based shortterm intervention for participants suffering from loneliness.

DETAILED DESCRIPTION:
Loneliness has a high prevalence in Western societies and poses a significant health problem. Among its many implications, loneliness has been associated with increased risk for coronary heart disease and stroke, depression, cognitive decline, dementia, and mortality. At the neural level, several networks may be involved in loneliness, including the reward circuitry, which mediates social reward, and the amygdala, which signals social threat. Intranasal OT has been reported to regulate activity in both the reward system and the amygdala. Therefore, it may serve as an adjunct to a cognitive-behavioral short-term intervention for high lonely participants.

In this randomized, double-blind, placebo-controlled design study, effects of intranasal OT (24 international units (UI)) as a pharmacological augmentation given before the start of four sessions of a cognitive-behavioral short-term intervention in groups of six to eight participants (based on established interpersonal psychotherapy modules to reduce loneliness) will be investigated. Healthy, but high lonely participants will complete functional magnetic resonance imaging (fMRI) tasks in a separate testing session before the start of the intervention (testing session 1). In the first session of the intervention, the psychotherapist will inform the participants about the procedure of the intervention and participants will get to know the other participants in their intervention group (testing session 2). In the next four sessions (testing sessions 3-6), participants will receive 24 IU of intranasal OT 30 minutes before the start of the intervention. Sessions of the intervention will be conducted weekly. After completion of the intervention, participants will again undergo fMRI scanning (testing session 7). Three weeks and three months after completion of the intervention, follow-up measurements of the experienced loneliness and subjective well-being will be collected.

All fMRI testing sessions (1 and 7) will include following tasks:

1. Blood-oxygen-level dependent (BOLD) signal will be measured while participants play a single-round trust game in the role of an investor. Participants will have to decide the amount of money they want to invest in an unknown trustee without receiving feedback about the decisions of the trustees. If the participant chooses to invest, that amount will be tripled and added to the trustee's account. The trustee may keep all of the money for him/herself or share the money with the investor. Participants will be informed of the collection of the trustee's decisions in a previous study for all possible investments. Furthermore, participants will view an image of a randomly chosen trustee from the previous study during the MRI session. In a control condition, participants will play a risk game and invest money in a computer (which will randomly decide whether the money will be shared).
2. BOLD signal will be assessed while participants undergo a social touch task. Trials will include slow (~ 5 cm/s) and fast touch (~ 20 cm/s) across 20 cm of the shins as well as a control condition (no touch). The touch will be administered by an experimenter that cannot be seen by the participants. After each trial, participants will be asked to rate the perceived comfort of the stimulation.

ELIGIBILITY:
Inclusion Criteria:

* UCLA loneliness scale score equal to or greater than 55

Exclusion Criteria:

* current psychiatric illness
* current psychiatric medication or psychotherapy
* MRI contraindication (e.g. metal in body, claustrophobia)
* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-09-26 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Scores on the UCLA Loneliness Scale | Five to seven weeks (+ Follow-Up measurements 3 weeks and 3 months after completion of the intervention)
  Loneliness, as measured via the University of California, Los Angeles (UCLA) loneliness scale before the start (testing session 1) and after completion of the intervention (testing session 7) (+ follow-up measurements 3 weeks and 3 months after completion of the intervention), will be analyzed using mixed ANOVAs with the software SPSS and Bonferroni-corrected post-hoc t-tests.
State loneliness (numeric rating scale) | Five to seven weeks (+ Follow-Up measurements 3 weeks and 3 months after completion of the intervention)
  State loneliness will be measured on a numeric rating scale ranging from 1 to 100 at the start and the end of each testing session and analyzed using mixed ANOVAs in SPSS and Bonferroni-corrected post-hoc t-tests.
Scores on the World Health Organization (WHO) Five Well-Being Index | Five to seven weeks (+ Follow-Up measurements 3 weeks and 3 months after completion of the intervention)
  Psychological well-being will be assessed using the World Health Organization (WHO) Five Well-Being Index before each testing session and analyzed using mixed ANOVAs in SPSS and Bonferroni-corrected post-hoc t-tests.
Scores on the Perceived Stress Scale | Five to seven weeks (+ Follow-Up measurements 3 weeks and 3 months after completion of the intervention)
  Perceived stress will be assessed using the Perceived Stress Scale (PSS-10) before each testing session and analyzed using mixed ANOVAs in SPSS and Bonferroni-corrected post-hoc t-tests.
Neural responses in the trust game | Five to seven weeks (fMRI task will be completed before the start and after the completion of the intervention and will take about 15 minutes)
  The BOLD signal as response to the trust game will be compared to the risk game and changes in the signal from testing session 1 to 7 will be compared between the OT and PLC groups. Results from both fMRI testing sessions will be compared to a non-lonely healthy control group (data were collected in a previous study with the same fMRI tasks in two fMRI sessions five to seven weeks apart from each other). Analyses will focus on anatomically defined regions of interests (ROIs) associated with trust (insula, amygdala, nucleus accumbens, and ventromedial prefrontal cortex). For analyses of fMRI data, standard procedures of the software SPM12 will be used. The family-wise error rate will be used to correct p-values for multiple comparisons and p < .05 will be considered significant. fMRI data will be correlated with behavioral data of the trust game and the UCLA Loneliness scores.
Amount of invested money in the trust game as an economic value of trust | Five to seven weeks (fMRI task will be completed before the start and after the completion of the intervention and will take about 15 minutes)
  Behavioral data of the trust game (invested money) will be analyzed using mixed ANOVAs in SPSS and compared between the OT and PLC groups. Post-hoc t-tests will be Bonferroni-corrected. Behavioral data will be correlated with fMRI data of the trust game and the UCLA Loneliness scores.
Neural responses to interpersonal touch | Five to seven weeks (fMRI task will be completed before the start and after the completion of the intervention and will take about 15 minutes)
  BOLD signals of slow touch trials will be contrasted with fast touch trials. Again, results of the OT group will be compared with the PLC group and results of lonely participants will be compared to the results of a non-lonely healthy control group. Analyses will focus on ROIs associated with the processing of social touch (amygdala, hippocampus, insula, and primary somatosensory cortex). For analyses of fMRI data, standard procedures of SPM12 will be used (preprocessing & a two-stage approach based on the general linear model for statistical analyses). The family-wise error rate will be used to correct p-values for multiple comparisons and p < .05 will be considered significant. Post-hoc t-tests will be Bonferroni-corrected. fMRI data will be correlated with behavioral data of the touch task and the UCLA loneliness scores.
Comfort ratings of interpersonal touch in the fMRI task (visual analogue scale) | Five to seven weeks (fMRI task will be completed before the start and after the completion of the intervention and will take about 15 minutes)
  Behavioral data of the fMRI interpersonal touch task (comfort ratings on a visual analogue scale) will be analyzed using mixed ANOVAs in SPSS and compared between the OT and the PLC group. Post-hoc t-tests will be Bonferroni-corrected. Comfort ratings will be correlated with fMRI data of the interpersonal touch task and the UCLA loneliness scores.
Therapeutic relationship (positive bonding) measured by the Group Questionnaire (GQ-D) | Five weeks
  The therapeutic relationship (positive bonding) will be measured after all intervention sessions using the Group Questionnaire (GQ-D; subscale Positive Bonding). OT effects will be analyzed by conducting mixed ANOVAs and Bonferroni-corrected post-hoc t-tests in SPSS.
Therapeutic relationship (positive working) measured by the Group Questionnaire (GQ-D) | Five weeks
  The therapeutic relationship (positive working) will be measured after all intervention sessions using the GQ-D (subscale Positive Working). OT effects will be analyzed by conducting mixed ANOVAs and Bonferroni-corrected post-hoc t-tests in SPSS.
Therapeutic relationship (negative relationship) measured by the Group Questionnaire (GQ-D) | Five weeks
  The therapeutic relationship (negative relationship) will be measured after all intervention sessions using the GQ-D (subscale Negative Relationship). OT effects will be analyzed by conducting mixed ANOVAs and Bonferroni-corrected post-hoc t-tests in SPSS.

SECONDARY OUTCOMES:
Interpersonal distance | Five to seven weeks (before the start and after the completion of the intervention)
  Interpersonal distance will be assessed by an adapted version of an established stop-distance paradigm. Participants start from a distance of ~ 2 m and move towards the investigator until their ideal distance is reached (trials 1 and 3) or until they feel slightly uncomfortable (trials 2 and 4). The task will be applied by the same investigator at testing sessions 1 and 7. Data will be analyzed using mixed ANOVAs and Bonferroni-corrected t-tests in SPSS to compare treatment group as well as lonely participants and non-lonely controls.
Neural activity at resting state | Five to seven weeks (fMRI task will be completed before start and after completion of the intervention and will take about 6 minutes)
  fMRI will be performed to measure BOLD-signal while participants lay in the MRI-scanner with eyes open. Participants will be instructed to look at a fixation cross for ~ 6 minutes. Functional connectivity will be analyzed using default preprocessing parameters implemented in the CONN-toolbox. Changes in functional connectivity will be contrasted between treatment groups and activity will be compared to those of non-lonely controls.

OTHER OUTCOMES:
Oxytocin plasma concentrations | Five to seven weeks (before the start and after the completion of the intervention)
  Oxytocin plasma concentrations will be assessed in testing sessions 1 and 7 before the fMRI scans will be conducted.

CONTACTS AND LOCATIONS:
Overall Officials: Rene Hurlemann, MSc, MD, PhD, Principal Investigator — University of Oldenburg
Locations (1):
- Department of Psychiatry, University of Bonn, Bonn, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Neuromodulation of Emotion (NEMO) research group — http://renehurlemann.squarespace.com/welcome/